CLINICAL TRIAL: NCT06123637
Title: Comparison of Analgesia Nociception Index-guided Anesthesia and Standard Anesthesia on Remifentanil Requirement in Desflurane Anesthesia
Brief Title: Analgesia Nociception Index-guided Anesthesia and Standard Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Ji Eun Kim, Assistant professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AJOUIRB-IV-2023-389
Record Dates: First submitted 2023-11-01; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesia nociception index group (Experimental)
  Interventions: Behavioral: Analgesia nociception index-guided anesthesia
- Standard group (Placebo Comparator)
  Interventions: Behavioral: Standard anesthesia

INTERVENTIONS:
Behavioral: Analgesia nociception index-guided anesthesia — Maintaining the blood pressure based on analgesia nociception index of >50 value
  Arms: Analgesia nociception index group
Behavioral: Standard anesthesia — Maintaining the blood pressure based on anesthesiologist's decision
  Arms: Standard group

SUMMARY:
The primary purpose of this study is to compare the analgesia nociception index-guided anesthesia and standard anesthesia on remifentanil requirement in desflurane anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gastric cancer

Exclusion Criteria:

* Conversion to open laparotomy
* Prior opioid abuse
* Prior infection
* Cardiac arrythmia

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Remifentanil requirement | at time of the end of skin suture (up to 4 hours)
  Assessing the total dose of remifentanil administered from skin incision until skin suture